CLINICAL TRIAL: NCT03330925
Title: Safety and Feasibility of the ElastiMed's SACS - Smart Active Compression Stocking
Brief Title: Safety and Feasibility of the ElastiMed's SACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElastiMed ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-001
Record Dates: First submitted 2017-10-25; First posted 2017-11-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-08

CONDITIONS: Compression; Vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ElastiMed's SACS (Experimental): Healthy Subjects which the Elastimed's SACS will be tried on
  Interventions: Device: ElastiMed's SACS

INTERVENTIONS:
Device: ElastiMed's SACS — A wearable medical device that improve circulation using smart materials

SUMMARY:
The main objective of this study is to demonstrate the safety and the feasibility of this device, and its ability to increase venous blood flow

Primary safety Endpoint:

To demonstrate the safety of the device- no serious adverse effect

Primary feasibility Endpoint:

Increase the blood flow velocity

The blood flow will be detected by a Duplex Ultrasonography test at the popliteal vein and the femoral vein.

The volunteers will rest at controlled environment room . Measurements will be performed after 30 min of rest without the device on the leg (baseline) and after 30 min of device activity .

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18<x<70 Years
2. Written informed consent has been sign by subject
3. With two healthy limbs - Normal blood flow according to leg deep vein Duplex test

Exclusion Criteria:

1. Positive pregnancy test
2. Breastfeeding woman
3. BMI 18.5 > X or X>25
4. Suffering from edema
5. Atrial fibrillation
6. DVT
7. Ulcers or cellulitis in regions covered by the compression device
8. Active phlebitis
9. Muscular disorders, or compartment syndrome
10. Heavy smoker >10 cigarettes a day
11. Subjects with altered mental status/inability to provide informed consent
12. Hematological disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Safety measured by the number of subjects with serious adverse events | 60 min
  The safety analysis set will contain of all subjects who were enrolled into the study.
  Individual listings of adverse events including type of device, adverse events (reported term), seriousness, duration, relationship to the study device, severity and the adverse events outcome will be provided
Device feasibility measured by an increase in blood flow velocity | 60 min
  The primary feasibility assessment will be based on the ability of the device to increase the blood flow velocity at the popliteal vein. The blood flow will be detected by a Duplex Ultrasonography test at the popliteal vein. Two Measurements will be performed, the first will be after 30 minutes of rest without the device on the leg (baseline) (T0) and the second will be after 30 min of device activity

CONTACTS AND LOCATIONS:
Overall Officials: Vered Shuster, PhD, Study Chair — ElastiMed ltd
Locations (1):
- Vascular Surgery Department, HILLEL YAFFE Medical Center,, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No